CLINICAL TRIAL: NCT02382536
Title: Infusion Pressure Delivering Insulin Diluent - BD's Scarlett vs. Medtronic's (MDT) Quickset in Healthy Adults
Brief Title: Monitoring the Infusion Pressure in Insulin Infusion Sets in Healthy Adults
Status: Completed | Type: Observational
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: DBC-14SCARL06
Record Dates: First submitted 2015-02-27; First posted 2015-03-06 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Diabetes
Keywords: Diabetes; Insulin therapy; insulin pump; Infusion sets
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infusion set: Each subject will receive a total of 4 simultaneous subcutaneous infusions of insulin diluent, two using the investigational device (BD Scarlett Infusion Set) and two using the the comparator (Medtronic QuickSet Infusion Set).
  Interventions: Device: BD Scarlett Infusion set; Device: Medtronic QuickSet Infusion Set

INTERVENTIONS:
Device: BD Scarlett Infusion set — Each subject will receive subcutaneous infusion from two investigational BD Scarlet infusion sets simultaneously, using a commercially available insulin pump to deliver insulin diluent (placebo) into the abdomen. Each infusion will run for approximately 4 1/2 hours.
Device: Medtronic QuickSet Infusion Set — Each subject will receive subcutaneous infusion from two Medtronic infusion sets simultaneously, using a commercially available insulin pump to deliver insulin diluent (placebo) into the abdomen. Each infusion will run for approximately 4 1/2 hours.

SUMMARY:
The purpose of this study is to compare the in-line fluid pressure (pressure of the fluid going through the tubing) and leakage (observation of fluid on and around the device) during and after subcutaneous infusion using two types of infusion sets. One infusion set is investigational, developed by BD, and the other is the Quick-set (Medtronic), which is commercially available. These infusion sets will be used with a commercially available insulin pump to deliver insulin diluent (an inactive liquid with no medication) for approximately 4 1/2 hours. During this time pressure and leakage will be continuously monitored.

DETAILED DESCRIPTION:
This is a single center, open label study.

Each subject is to receive up to 4 basal/bolus diluent infusions in the abdomen with the BD Scarlett and the Medtronic Quick-set®; 2 Scarlett infusion sets and 2 Quick-set infusion sets. The order of device placement will be randomized.

After insertion, insulin diluent will be delivered at a rate of 0.01 mL/hour (equivalent in volume and rate to 1.0 unit/hour of U-100 insulin) via the insulin pump for a minimum of 3 hours. After 3 hours of basal infusion, a bolus of 0.1 mL (equivalent to 10 units) will be delivered via the insulin pump and basal infusion continued for a minimum of 1 additional hour.

At the end of the final basal infusion period, the infusion set tubing will be clamped to mimic an occlusion event and allowed to run until either an occlusion alert ("no delivery") is signaled by the pump, or a minimum of 30 minutes, whichever comes first. Infusion pressure data will be collected during the entire infusion period, including the time the tubing is clamped. After removal of the device from the body, the presence of fluid on the application site skin (Leakage) will be determined by visual assessment then measured using gravimetric analysis, if applicable.

ELIGIBILITY:
Inclusion Criteria:

1. Must be between the ages of 18-75 years of age (inclusive)
2. In stable health status with no acute or significant illness, in the opinion of the investigator.
3. Able to read, write and follow study instructions in English.
4. Able and willing to provide informed consent.
5. Able and willing to complete all study procedures.

Exclusion Criteria:

1. Pregnant (self-attestation)
2. BMI > 35
3. Currently taking anti-platelet therapy or anticoagulants (Use of up to 81 mg per day of aspirin is permitted)
4. History of bleeding disorder or easy bruising
5. Known blood borne infections
6. Diabetes on insulin therapy
7. History of recurrent dermatological condition or skin disorder (e.g. psoriasis, eczema)
8. Gross skin anomalies and abnormalities (e.g. scars, stretch marks, discolorations, tattoos, superficial masses, other) located at or very close to the intended infusion sites on the abdomen
9. Subjects with excessive hair on the abdomen who are unwilling to have excessive hair removed by Site Staff
10. Fear of needles, history of symptomatic low blood pressure or history of fainting (syncope) during hypodermic injections
11. History of allergic reaction to adhesives, metals, latex, or plastics.
12. Any other condition the PI or designee deems to pose a risk to the subject in the study.
13. Currently participating in any other clinical investigation that conflicts with this one, or who have participated in a study with the same indication within the prior 30 days that the Principal Investigator or designee believes will conflict with outcomes or ability of the subject to complete all activities required in this study.
14. Employed by, or currently serving as a contractor or consultant to BD

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
In-line fluid pressure | Continuous measure for 4-5 hours after insertion
  Infusion pressure profiles will be measured by an inline pressure transducer and recorded by a data logger. Pressure profiles will be evaluated by type of infusion set. The occurrence of pressure events (continuous pressure rises or flow interruptions of at least 30 minutes) will be assessed.

SECONDARY OUTCOMES:
Leakage | Immediately upon device removal
  Upon removal of the infusion set, the infusion site and device will be checked for fluid leakage. If leakage is observed, the infusion site device hub/skin interface will be swabbed for fluid with a pre-weighed swab. The swab will be re-weighed to determine the amount of fluid. Fluid collected at infusion site and the device/skin interface will not be classified as leakage if the measured volume is less than 0.005 mL (equivalent to 0.5 units U-100 insulin).

OTHER OUTCOMES:
Number of subjects with adverse events | Approximately 6 hours from device application until study completion.
  During the study visit subjects will be asked about adverse events that may have occurred. All adverse events, e.g. skin irritation, allergic reaction, excessive pain, will be evaluated, appropriately treated and followed up as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Phillip LaStella, MD, Principal Investigator — TKL Research
Locations (1):
- TKL Research, Fair Lawn, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No